CLINICAL TRIAL: NCT07400016
Title: Efficacy of Superoxide Dismutase Spray in Preventing Radiation Dermatitis in Patients With Head and Neck Cancer .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HX2024-134-5
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A placebo spray (Placebo Comparator): A placebo spray containing excipients (lactose, potassium sorbate, and sorbitol) in addition to no SOD.
  Interventions: Other: Placebo Spray
- Superoxide dismutase (SOD) Spray (Experimental)
  Interventions: Other: SOD spray

INTERVENTIONS:
Other: Placebo Spray — Patients are instructed to apply the placebo spray to the treatment area twice daily, starting three days before radiotherapy (RT) and continuing until two weeks after treatment completion. The spray should be used to cover the entire treatment area. Patients are also advised not to use the spray within four hours before RT. They are required to keep the skin in the radiotherapy area dry and clean and to refrain from using other topical agents in the irradiated area. Use of the spray should be discontinued if dermatitis of grade 2 or higher occurs.
  Arms: A placebo spray
Other: SOD spray — Patients are instructed to apply a thin layer of SOD spray to the treatment area twice daily, beginning three days before radiotherapy (RT) and continuing- Page 3 of 6 Arms Assigned Interventions until two weeks after treatment completion. The application should cover the entire treatment area. Patients are also advised not to use the spray within four hours before RT to avoid potential buildup effects. They are required to keep the skin in the radiotherapy area dry and clean and to refrain from using other topical agents in the irradiated area. Use of the spray should be discontinued if dermatitis of grade 2 or higher occurs.
  Arms: Superoxide dismutase (SOD) Spray

SUMMARY:
Radiotherapy always results in many complications such as radiation dermatitis,dry mouth, cranial nerve damage, and swallowing function. Among them,radiation dermatitis is confirmed to occur in the majority of tumor patientsreceiving radiotherapy, which not only affects the appearance but also causesthe interruption of radiotherapy in severe cases. At present, there is no standard treatment for radiation dermatitis. Superoxide dismutase (SOD) Spray is able to removefree radicals produced during radiotherapy, which may provide a new way andmethod for the prevention and treatment of radiation dermatitis. In addition,the product has obtained a safety assessment report from a third-party testingorganization, proving that it has fully met the applied human body standards. This clinical trial studies the effect of superoxide dismutase (SOD) Spray in preventing radiationdermatitis in Head and Neck Cancer.

DETAILED DESCRIPTION:
Radiotherapy is an essential modality in the curative and palliative management of head and neck malignancies, but it is frequently accompanied by a spectrum of acute and late toxicities, including radiation dermatitis, xerostomia, cranial nerve injury, and dysphagia. Radiation dermatitis, an inflammatory skin reaction to ionizing radiation, develops in the majority of patients undergoing external beam radiotherapy to the head and neck region and ranges from mild erythema and dry desquamation to moist desquamation and ulceration in severe cases. Clinically significant skin injury not only compromises patients' quality of life through pain, pruritus and cosmetic disfigurement, but may also necessitate treatment interruptions or dose reductions, which have been associated with inferior tumor control and survival outcomes in several studies. The pathophysiology of radiation dermatitis is multifactorial and involves direct radiation-induced DNA damage, endothelial cell injury, cytokine-mediated inflammatory cascades, and generation of reactive oxygen species (ROS). ROS, particularly superoxide anions, play a central role in propagating oxidative stress, lipid peroxidation and subsequent tissue injury. Current management strategies for radiation dermatitis are largely supportive and empirical, including skin hygiene measures, topical corticosteroids, emollients, dressings for moist desquamation, and pain control; however, there is no universally accepted standard of care and robust high-quality evidence for many interventions remains limited. Antioxidant-based topical and topical-delivery agents have been explored as prophylactic and therapeutic options to mitigate radiation-induced skin injury by neutralizing ROS and modulating inflammatory responses. Superoxide dismutase (SOD) is a key endogenous antioxidant enzyme that catalyzes the dismutation of superoxide radicals into oxygen and hydrogen peroxide, thereby reducing oxidative stress. Preclinical studies and early clinical reports suggest that SOD-containing formulations or SOD-mimetic compounds can decrease markers of oxidative damage, attenuate inflammatory signaling, and reduce histologic evidence of radiation-induced dermal injury. The investigational SOD spray evaluated in this trial is formulated for topical aerosolized delivery to irradiated skin surfaces, which may offer advantages in ease of application, uniform coverage of complex anatomical regions in the head and neck, and patient compliance compared with creams. Early-phase studies of topical sprays delivering antioxidants or SOD-mimetic agents have- Page 2 of 6 demonstrated favorable tolerability and potential reductions in the severity of acute radiation dermatitis, though data remain limited and heterogeneous. The SOD spray in this study has undergone third-party safety assessment and meets human-use standards, supporting its tolerability for topical application. Given the biological plausibility, encouraging preliminary data for antioxidant approaches, and the unmet clinical need for effective prophylaxis against radiation dermatitis, this randomized clinical trial aims to evaluate the efficacy and safety of SOD spray in preventing radiation dermatitis among patients with head and neck cancer undergoing definitive or adjuvant radiotherapy. Primary endpoints include incidence and maximal grade of acute radiation dermatitis based on standardized scoring systems, while secondary endpoints will assess time to onset, patient-reported skin symptoms and quality of life, treatment interruptions, and safety/tolerability metrics. The trial's findings may inform evidence-based recommendations for topical antioxidant prophylaxis in the radiotherapy setting and potentially improve treatment adherence and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
* 2. Patients considered candidates for high-dose RT either as primary treatment or as postoperative treatment after surgical resection and patients planned to receive concomitant boost fractionation or concurrent systemic chemotherapy

Exclusion Criteria:

* 1. Eastern Cooperative Oncology Group performance status of #2;
* 2.Pre-existing skin rash, ulceration or open wound in the treatment area;
* 3. Known allergy to trolamine or fullerene;
* 4. Inflammatory or connectivetissue disorder of the skin;
* 5. History of head and neck radiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 2 or higher radiation dermatitis. | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Patients are assessed weekly for radiation dermatitis by an experienced radiation oncology nurse according to the Radiation Therapy Oncology Group (RTOG) scale. The RTOG scale categorizes acute skin toxicity into grades 0-4, with the higher the grade the more severe the patient's acute radiation dermatitis. Grade 0 means no change over baseline. Grade 1 means follicular, faint, or dull erythema; epilation, dry desquamation, or decrease in sweating. Grade 2 means tender, bright erythema; patchy, moist desquamation or moderate edema. Grade 3 means confluent, moist desquamation other than skin folds; pitting edema. Grade 4 means ulceration, hemorrhage, necrosis.

SECONDARY OUTCOMES:
The time to onset of grade 2 or higher radiation dermatitis. | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Time from the first day of radiotherapy to the first determination of grade 2 or higher radiation dermatitis.
The duration of grade 2 or higher radiation dermatitis. | From the start of radiotherapy to 4 weeks after completion of radiotherapy.
  The first determination of grade 2 or higher radiation dermatitis to the first instance of grade 1 or 0 radiation dermatitis, without a subsequent instance of grade 2 or higher radiation dermatitis. Patients without observed grade 2 or higher radiation dermatitis were assigned a duration of 0 days.
The maximum skin toxicity. | From the start of radiotherapy to 4 weeks after completion of radiotherapy.
  The maximum grade of RTOG skin toxicity between 0 and 4.
The Skindex-16 instrument. | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  The Skindex-16 is a commonly used tool to measure the effect of skin diseases on the QoL of patients. Skindex-16 consists of domain scores that assess how symptoms, emotions, and functioning from the skin issue affect the QOL of patients with acne. The overall score averages the 3 domain scores, all of which are normalized to a 0 to 100 scale, where 0 indicates that their skin condition has no impact on QOL and 100 represents maximal impact on QOL for the worse.
EORTC QLQ-C30. | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  The EORTC QLQ-C30 consists of five functional scales, nine symptom scales and one global quality of life (QoL) scale, and has been validated in an international setting.The questionnaire uses a four-point Likert scale to indicate the extent of problems experienced, ranging from 'not at all' to 'very much'. The answers for each domain are converted to a score ranging from 0 to 100#or functional scales, high scores represent a high level of QoL#and for symptom scales high scores indicate a poor QoL.
EORTC QLQ-H&N35 | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  The EORTC QLQ-H&N35 covers issues specific to HNC patients and includes 18 symptom scales; it has been validated in an international setting and is used extensively in HRQoL research. The questionnaire uses a four-point- Page 4 of 6 Likert scale to indicate the extent of problems experienced, ranging from 'not at all' to 'very much'. The answers for each domain are converted to a score ranging from 0 to 100#or functional scales, high scores represent a high level of QoL#and for symptom scales high scores indicate a poor QoL.
Adverse events. | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version.

IPD SHARING:
Plan to Share IPD: No